CLINICAL TRIAL: NCT06807060
Title: A Municipality Implemented Behavioural Intervention to Improve Quality of Life Among Older Adults: Protocol for a Mixed-Methods Pilot Case Study
Brief Title: A Municipality Implemented Behavioural Intervention to Improve Quality of Life Among Older Adults
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lund University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2024-01607-01
Record Dates: First submitted 2025-01-24; First posted 2025-02-04 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Quality of Life
Keywords: Complex intervention; Behavioural change; Environmental proactivity; Older adults; Usability; Quality of Life; Daytime outdoor walking
MeSH Terms: interventions — Light; Exercise; Sleep

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): All participants receive the same intervention, including noninvasive approaches (both education and behavioural).
  Interventions: Behavioral: 'Light, activity and sleep in my daily life' intervention

INTERVENTIONS:
Behavioral: 'Light, activity and sleep in my daily life' intervention — The intervention is complex in that it considers multiple factors (e.g., light-related behaviour, physical activity and sleep behaviour) and multiple components (e.g., cognitive goal setting and implementation).
  The intervention is delivered as a web-based course on a digital learning platform. Course material is placed in nine modules covering electric lighting, daylight, physical activity outdoors and sleep. Besides online material, the course includes a test kit containing light bulbs, a sleep mask, a checklist for the room inventory, a cap, a notebook, and a sleep diary. The purpose of the test kit is to encourage experimentation and provide handouts and printed copies to facilitate the completion of assignments.

SUMMARY:
Ageing is associated with circadian rhythm sleep disorders, poor sleep at night, less physical activity and more time spent indoors, affecting the wellbeing of older adults. Their sleep and mood could benefit from daytime outdoor physical activity, exposure to daylight, better indoor lighting and sleep routines. However, maintaining or increasing one's physical activity can be challenging depending on individual behavioural conditions, e.g., having the physical and cognitive capacity (capability), finding the activity enjoyable and relevant to one's needs (motivation), and having a supportive social and physical environment (opportunity), such as a walk-friendly environment. To address these challenges, a complex behavioural intervention was developed. The intervention is delivered as a web-based course ('Light, activity and sleep in my daily life', LAS) that targets light-related behaviour, outdoor walking and sleep behaviour among community-dwelling older adults. This protocol describes a pilot case study aiming to evaluate the usability and usefulness of the LAS intervention, the intervention outcomes and whether changes to routines are sustained.

Eligible intervention participants (target N=40) are Swedish-speaking adults (≥ 70 years), living in one-person households in apartments in four municipalities. Participants complete questionnaires assessing intervention outcome measures (e.g., quality of life), are interviewed about their daily routines, and wear an accelerometer which tracks activity and rest at the baseline. Participants then enrol in a 9-week course, including self-studies at home and four physical meetings at the senior citizen meeting point. Baseline measures are repeated after the course, at 3, 6 and 10 months after baseline. In addition, participants evaluate the intervention's usability and usefulness after the course at 3 months and are interviewed at 6 months after baseline about perceived enablers and inhibitors to daytime outdoor walking.

Results will inform a subsequent larger case study focused on optimising the LAS intervention's content and delivery procedures to enable an intervention better integrated into municipal health promotion services/strategies. An anticipated long-term outcome is continued active ageing and independence.

DETAILED DESCRIPTION:
Development of the intervention: 'Light, activity and sleep in my daily life' The 'Light, activity and sleep in my daily life' (LAS) intervention directed at older adults was developed to promote wellbeing through increased physical activity, enhanced mood and sleep, and improved lighting and darkness conditions at home. The intervention focuses on health promotion through changes to routines (light-related behaviour, outdoor physical activity and sleep behaviour) and environmental proactivity. The latter refers to persons who modify their environments to live a healthy and independent life. Environmental modifications include interior lighting, filtering daylight and blocking light at night, without risking accidents when getting up at night, and furniture arrangement.

The intervention is complex in that it considers multiple factors (e.g., light-related behaviour, physical activity and sleep behaviour) and components (e.g., cognitive goal setting and implementation. The intervention addresses self-identified needs, which can make it more effective.

The intervention is delivered as a web-based course on a digital platform and includes one introductory physical meeting and three additional physical meetings. Course material is placed in nine modules covering electric lighting, daylight, physical activity outdoors and sleep. Each completed module ends with a brief online evaluation. Besides online material, the course includes a test kit containing light bulbs, a sleep mask, a checklist for the room inventory, a cap, a notebook, and a sleep diary. The purpose of the test kit is to encourage experimentation and provide handouts and printed copies to facilitate the completion of assignments.

In 2021-2022 usability evaluations of a first version were conducted in a full-scale model of an apartment by two sets of participants: in a first round by experts and in a second round by pensioners representing the target users (community-dwelling adults aged 70 and over). Intervention content and design features were refined based on their feedback. In autumn 2022, intervention usability and study feasibility were evaluated in real-world homes by eight participants aged 71-84 (27). The conclusion was that only minor changes to the intervention were needed based on participants' feedback. Regarding the locality for the physical meetings, the researchers found the municipality's senior citizen meeting point suitable for the purpose, and participants appreciated that meetings were at the same place. One finding was the need to extend the time for recruitment, and advertising in the local newspapers should be considered to reach a wider group of potential volunteers.

Based on the study findings from the field, the following design changes were made to the online intervention content: the weekly evaluation form was revised so intervention participants can provide textual feedback to the course leader/interventionist; instructions for downloading the light meter app to the phone were revised; and text links were updated.

This pilot case study aims to evaluate the usability and acceptance of the LAS intervention, the intervention outcomes and whether changes to routines are sustained. In addition, perceived enablers and inhibitors to daytime outdoor walking will be identified.

The primary objectives are as follows:

1. To evaluate the usability and usefulness of the intervention, that is, determine if the online intervention content is easy to use and the intervention is useful for older adults 70 and over.
2. To evaluate the acceptance of intervention delivery procedures (locality of physical meetings, recruitment) to municipal staff (potential service providers).
3. To identify motivation/capabilities/opportunities relating to outdoor physical activity (e.g., perceived enablers and inhibitors to daytime outdoor walking).
4. To develop further training material for future course leaders/interventionists in dialogue with the municipal partners.

A secondary objective is to gain insight into the potential effectiveness of the intervention in terms of activity and rest patterns, mood, sleep quality, behavioural skills and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* aged 70 and over, ambulatory and sighted,
* Swedish speaking,
* living independently in one-person households in ordinary apartments and
* receiving no or limited home care services.

Exclusion Criteria:

Study participants will be excluded if they have any condition that makes it difficult to participate.

Min Age: 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-05-15 (Actual); Primary Completion 2026-10-16 (Estimated); Study Completion 2026-10-16 (Estimated)

PRIMARY OUTCOMES:
Usability | At one timepoint: 3 months after baseline
  System Usability Scale score. The usability of the intervention, that is, if the online content is easy for the intervention participants to use, will be evaluated through a usability testing questionnaire (perceptions of complexity, integration of functions, consistency). Following published instructions on scoring of the 10-item System Usability Scale (SUS), a total usability score will be calculated ranging from 0 to 100. Higher SUS scores indicate greater usability. Based on empirical evaluations of the SUS, a SUS score below 50 indicates usability difficulties, while scores in the 70s and 80s are considered promising.

SECONDARY OUTCOMES:
Mood | At four timepoints: baseline, 3, 6 and 13 months after baseline
  Short Swedish Core Affect Scales. Two scales measuring two dimensions, 'valence' (including three adjective pairs) and 'activation' (including three adjective pairs). Scores for each dimension can range from 1 to 9, with higher scores indicating better mood.
Sleep quality | At four timepoints: baseline, 3, 6 and 13 months after baseline
  Sleep Disturbance instrument, Patient-Reported Outcomes Measurement Information System (PROMIS) Bank v1.0. Assessing sleep disturbance, including four items. The total raw score can range from 32 to 73.3, with higher scores indicating worse sleep quality.
Behavioural skill | At four timepoints: baseline, 3, 6 and 13 months after baseline
  A New General Self-efficacy Scale. Assessing general self-efficacy, including eight items (goal achievement, task accomplishment, obtaining important outcomes, succeeding at most any endeavour, overcoming challenges, effective performance, doing tasks well, performing well even when things are tough). The global score can range from 1 to 5, with higher scores indicating higher self-efficacy.
Quality of life | At four timepoints: baseline, 3, 6 and 13 months after baseline
  World Health Organization Quality of Life (BREF) questionnaire. Assessing quality of life over four domains (physical health, psychological, social relationships, environment). Scores for each domain can range from zero to 100, with higher scores indicating better quality of life.
Sleep (activity and rest patterns) | At four timepoints: baseline, 3, 6 and 13 months after baseline. Duration of time over which each participant is assessed: 7 days (not used during shower)
  Performance-based measure using a wrist-worn accelerometer (ActiGraph wGT3X-BT, ActiGraph LLC, Pensacola, FL)
Physical activity | At four timepoints: baseline, 3, 6 and 13 months after baseline. Duration of time over which each participant is assessed: 8 days (not used during shower)
  Performance-based measure using a wrist-worn accelerometer (ActiGraph wGT3X-BT, ActiGraph LLC, Pensacola, FL). Assessing light, moderate-to-vigorous and vigorous physical activity (minutes).
Sedentary behaviour | At four timepoints: baseline, 3, 6 and 13 months after baseline. Duration of time over which each participant is assessed: 7 days (not used during shower)
  Performance-based measure using a wrist-worn accelerometer (ActiGraph wGT3X-BT, ActiGraph LLC, Pensacola, FL). Assessing sedentary time (minutes).
Steps | At four timepoints: baseline, 3, 6 and 13 months after baseline. Duration of time over which each participant is assessed: 7 days (not used during shower)
  Performance-based measure using a wrist-worn accelerometer (ActiGraph wGT3X-BT, ActiGraph LLC, Pensacola, FL). Assessing the number of steps.

OTHER OUTCOMES:
Computer anxiety | At two timepoints: baseline and 3 months after baseline
  Short Computer Anxiety Scale. Assessing computer anxiety, including six items. The global score can range from 6 to 36, with higher scores indicating higher computer anxiety.
Lighting quality | At two timepoints: baseline and 3 months after baseline
  Perceived Indoor Lighting Quality. Five bipolar adjective scales measuring the dimension 'Strength' and five measuring the dimension 'Hedonic tone'. Scores for each dimension can range from 1 to 7, with higher scores indicating higher 'Strength' (perceived strength quality) and higher 'Hedonic tone' (perceived comfort quality).

CONTACTS AND LOCATIONS:
Locations (4):
- Sweden (4):
  - Gothenburg Municipality, Gothenburg
  - Jönköping Municipality, Jönköping
  - Lund Municipality, Lund
  - Malmö Municipality, Malmo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gerhardsson KM, Hassan M, Tornberg AB, Schmidt SM. Usability and feasibility of an online intervention for older adults to support changes to routines and the home ('Light, activity and sleep in my daily life'). BMC Public Health. 2024 Oct 14;24(1):2808. doi: 10.1186/s12889-024-20309-y. PMID 39402489